CLINICAL TRIAL: NCT00567697
Title: A Randomized Study Comparing the Safty Anf Efficacy of Ranibizumab (Lucentis®) to Sham in Patients With Macular Edema Secondary to Central Retinal Vein Occlusion (CRVO
Brief Title: A Randomized Study Comparing Ranibizumab to Sham in Patients With Macular Edema Secondary to CRVO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aleris Helse (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ROCC study 2007
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Central Retinal Vein Occlusion; Macular Edema
Keywords: ranibizumab; CRVO; macular edema; sham
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 0.5 ml 10mg/ml (0.5 mg) ranibizumab for intravitreal injection
  Interventions: Drug: ranibizumab
- B (Sham Comparator)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5 ml 10mg/ml (0.5 mg) ranibizumab for intravitreal injection. Monthly injection for 3 months, followed by reinjection if edema for a total of 6 months.
  Arms: A
Drug: ranibizumab — Sham injection with an empty, sterile 3-ml stopped glass vial. # monthly sham-injections, followed by reinjection for 3 months if present edema.
  Arms: B

SUMMARY:
A prospective multicenter study comparing patients with CRVO amd secondary macular edema treated with ranibizumab versus sham. Safety and efficacy will be evaluated. Patients will be randomized in a 1:1 ratio to one of the two arms. 32 patients, 6 months follow up. There will be monthly visits with injection the first three months and subsequently new injection if present edema.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 50 years
2. Patients who have findings consistent with CRVO
3. Patients who have a history of decreased visual acuity ≤ 6 months
4. Patients who have a best corrected visual acuity (BCVA) letter score in the study eye of ≤ 73 (4 m distance) or ≥ 6 (1 m distance) using an ETDRS chart
5. Patients who have a macular edema verified by OCT
6. Patients who have macular edema in the study eye with the following characteristics as determined by fluorescein angiography:

   * secondary to non-iscemic CRVO defined as non-perfusion < 10 DA OR
   * secondary to ischemic CRVO defined as non-perfusion > 10 DA
7. Willing and able to give written informed consent and who are willing and able to comply with study procedures
8. Ability to cooperate with photo and OCT examinations

Exclusion Criteria:

1. Neovascularisations in the study eye at baseline
2. Previous treatment with or participation in a clinical trial (for either eye) involving anti-angiogenics drugs
3. Use of other investigational drugs
4. Prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal laser photocoagulation, vitrectomy, or transpupillary thermotherapy.
5. History of submacular surgery in the study eye, glaucoma filtration, corneal transplantation surgery
6. Previous or current intravitreal or sub-Tenon drug delivery in the study eye
7. Laserphotocoagulation (juxtafoveal or extrafoveal) in the study eye within one month preceding Baseline
8. Extracapsular extraction of cataract with phacoemulcification within three months preceding Baseline, or a history of post-complications within the last 12 months preceding Baseline in the study eye (uveitis, cyclitis etc)
9. History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication)
10. Previous violation of the posterior capsule in the study eye unless it occurred as a result of YAG laser posterior capsulotomy in assosiation with prior, posterior chamber lens implantation
11. Afakia with absence of the posterior capsule in the study eye
12. Active intraocular inflammation in the study eye
13. Any active infection involving the ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as ideopathic or autoimmune-associated uveitis in either eye
14. Vitreous hemorrhage or history og rhegmatogenous retinal detachment or macular hole in the study eye
15. Any current intraocular condition in the study eye (cataract or diabetic retinopathia) that in the opinion of the investigator, could either require medical or surgical intervention during the study period for the next 6 months
16. Ocular condition that requires chronic concomitant therapy with systemic or topical ocular corticosteroids.
17. Current treatment for active systemic infection.
18. Current use or likely need for systemic medications known to be toxic to the lens, retina or optic nerve.
19. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or might affect interpretation of the results of the study or render the subject at high risk for treatment complications
20. History of hypersensitivity or allergy to fluorescein
21. Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed
22. Pregnant or nursing (lactating) women
23. Pre-menopausal women of child-bearing potential not using adequate contraception.
24. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrance or metastases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome measure is the mean change from baseline in BCVA score | 6 months

SECONDARY OUTCOMES:
Mean change from baseline in BCVA score, central foveal thickness and in the NEI VFQ-25 near activities subscale. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Kinge, MD DMSc, Principal Investigator — Aleris Helse, Oslo
Locations (4):
- Norway (4):
  - Bettina Kinge, Retinaklinikken Aleris, Oslo
  - Ingar Stene Johansen, Oslo
  - Vegard Forsaa, Stavanger
  - Kristian Fossen, Tromsø

REFERENCES:
- [Derived] Kinge B, Stordahl PB, Forsaa V, Fossen K, Haugstad M, Helgesen OH, Seland J, Stene-Johansen I. Efficacy of ranibizumab in patients with macular edema secondary to central retinal vein occlusion: results from the sham-controlled ROCC study. Am J Ophthalmol. 2010 Sep;150(3):310-4. doi: 10.1016/j.ajo.2010.03.028. Epub 2010 Jun 29. PMID 20591399